CLINICAL TRIAL: NCT01088620
Title: CHAMP - An Open-label, Randomised, Multicentre, Phase II Clinical Study of Panitumumab Plus Pemetrexed and Cisplatin (PemCisP) Versus PemCis in the First-line Treatment of Patients With Stage IIIB or IV Primary Nonsquamous Non-small Cell Lung Cancer, With Particular Regard to the KRAS Status
Brief Title: Panitumumab Plus Pemetrexed and Cisplatin (PemCisP) Versus PemCis in the First-line Treatment of Patients With Non-small Cell Lung Cancer
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: the DSMB stopped the trial due to unacceptable side effects in the experimental arm which has not yet been verified
Sponsor: WiSP Wissenschaftlicher Service Pharma GmbH (Other)
Collaborators: Gesellschaft fur Medizinische Innovation - Hamatologie und Onkologie mbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WISP_AG47; 2009-014677-41 (EudraCT Number); GMIHO-006/2008 (Other: GMIHO)
Record Dates: First submitted 2010-03-16; First posted 2010-03-17 (Estimated); Last update posted 2013-03-14 (Estimated); Status verified 2013-03

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: NSCLC; Stage IIIb or IV; Nonsquamous; KRAS-Wildtype
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Panitumumab; Pemetrexed; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Panitumumab plus pemetrexed and cisplatin (PemCisP) (Experimental)
  Interventions: Drug: Panitumumab; Drug: Pemetrexed; Drug: Cisplatin
- Pemetrexed and cisplatin (PemCis) (Active Comparator)
  Interventions: Drug: Pemetrexed; Drug: Cisplatin

INTERVENTIONS:
Drug: Panitumumab — Panitumumab 9 mg/kg BW will be administered IV every 3 weeks (q3w) for a maximum of four cycles.
  In case of CR, PR or SD status at the end of the combination treatment, a panitumumab single drug treatment, consisting of 9 mg/kg BW administered every 3 weeks, will be performed until detection of disease progression.
  Other Names: Vectibix
  Arms: Panitumumab plus pemetrexed and cisplatin (PemCisP)
Drug: Pemetrexed — Pemetrexed 500 mg/m² will be administered IV every 3 weeks (q3w) for a maximum of four cycles.
  Other Names: Alimta
Drug: Cisplatin — Cisplatin 75 mg/m² will be administered IV every 3 weeks (q3w) for a maximum of four cycles.

SUMMARY:
The purpose of this trial is to estimate the therapeutic efficacy of the experimental targeted regimen including the EGFR antibody panitumumab (in combination with pemetrexed and cisplatin) in relation to the standard combination in patients with a KRAS wild-type stage IIIB or IV primary nonsquamous non-small cell lung cancer. It is expected that the progression free survival rate at 6 months is improved by the targeted regimen.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of inoperable stage IIIB or IV primary pulmonary nonsquamous NSCLC (according to UICC staging valid until 2008)
* Sufficient representative sample material for KRAS analysis
* Wild-type KRAS
* Informed consent of the patient
* Aged at least 18 years
* WHO Performance Status 0-2
* At least one unidimensional, measurable tumour parameter according to RECIST
* Life expectancy of al least 12 weeks
* Adequate haematological, hepatic, renal and metabolic function parameters:

  * Leukocytes > 3000/mm³, ANC ≥ 1500/mm3, platelets ≥ 100,000/mm3, Creatinine clearance ≥ 50 ml/min and serum creatinine ≤ 1.5 x upper limit of normal
  * Bilirubin ≤ 1.5 x upper limit of normal, GOT-GPT ≤ 2.5 x upper limit of normal in absence of liver metastases, or ≤ 5 x upper limit of normal in presence of liver metastases, AP ≤ 5 x upper limit of normal
  * Magnesium ≥ lower limit of normal; calcium ≥ lower limit of normal

Exclusion Criteria:

* Prior chemotherapy
* Clinically manifest, uncontrolled brain metastases
* Prior radiotherapy of the parameters to be measured
* Peripheral neuropathy NCI grade > 1
* Subject pregnant or breast feeding, or planning to become pregnant within 6 months after the end of treatment.
* Subject (male or female) is not willing to use highly effective methods of contraception (per institutional standard) during treatment and for 6 months (male or female) after the end of treatment (adequate: oral contraceptives, intrauterine device or barrier method in conjunction with spermicidal jelly).
* Serious concurrent diseases.
* Major surgery within the last 4 weeks before recruitment
* On-treatment participation in a clinical study in the period 30 days prior to inclusion.
* Clinically significant cardiovascular disease in (incl. myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) ≤ 1 year before enrolment.
* Ongoing or active infection, including active tuberculosis or known infection with human immunodeficiency virus.
* Superior vena cava syndrome contraindicating hydration.
* History of interstitial lung disease, e.g. pneumonitis or pulmonary fibrosis or evidence of interstitial lung disease on baseline chest CT scan.
* Patient with mild to moderate renal insufficiency who are unable to interrupt salicylates (like aspirin) or other nonsteroidal anti-inflammatory drugs (NSAIDS) for a 5-day period starting 2 days before administration of pemetrexed (8-day period for long-acting agents such as piroxicam). Exception: Low dose aspirin (acetyl salicylic acid) intake up to 150 mg per day is permitted without interruption.
* Presence of clinically significant third-space fluid collections, for example, ascites or pleural effusions that cannot be controlled by drainage or other procedures
* Inability or unwillingness to take folic acid, vitamin B12 supplementation or dexamethasone (or equivalent corticosteroid); or any other inability to comply with protocol or study related procedures
* Prior or concurrent malignancy (≤ 5 years prior to enrolment in study) except non-melanoma skin cancer or cervical carcinoma FIGO stage 0-1 if the patient is continuously disease-free
* Known allergic reactions on study medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2010-04; Primary Completion 2013-01 (Actual); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival rate at 6 months | 6 months

SECONDARY OUTCOMES:
Determination of the tumour response | 6 months
Duration of response | 6 months
Overall survival | 6 month
Adverse effects / toxicity | 6 months
Quality of life assessment | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Schütte, MD, Principal Investigator — Krankenhaus Martha-Maria Halle-Dölau
Locations (20):
- Germany (20):
  - Schwerpunktpraxis für Hämatologie und Internistische Onkologie, Gesundheitszentrum St. Marien GmbH, Amberg
  - Universitätsklinikum Charité - Campus Mitte, Berlin
  - Charité Campus Benjamin Franklin Medizinische Klinik m. S. Hämatologie und Onkologie, Berlin
  - HELIOS Klinikum Emil von Behring - Lungenklinik Heckeshorn, Berlin
  - Augusta-Kranken-Anstalt gGmbH, Bochum
  - Johanniter-Krankenhaus Bonn, Bonn
  - Kliniken der Stadt Köln, Krankenhaus Merheim, Cologne
  - Carl-Thiem-Klinikum Cottbus gGmbH, Cottbus
  - Medizinische Fakultät Carl Gustav Carus der Technischen Universität Dresden Medizinische Klinik 1, Dresden
  - Katholisches Klinikum Duisburg/St. Johannes-Hospital, Duisburg
  - Klinikum Frankfurt (Oder) GmbH, Frankfurt (Oder)
  - Krankenhaus Großhansdorf GmbH Onkologischer Schwerpunkt, Großhansdorf
  - Krankenhaus - Martha-Maria Halle-Dölau GmbH, Halle
  - Universitätsklinikum Halle (Saale), Klinik und Poliklinik für Innere Medizin I, Halle
  - Universitätsklinikum Jena, Klinik für Innere Medizin I, Jena
  - Onkologische Schwerpunktpraxis Dr. Stauch, Kronach
  - UK-SH, Campus Lübeck, Med. Klinik III, Lübeck
  - LMU-Klinikum der Universität München, Medizinische Klinik München-Innenstadt, München
  - Oncologianova GmbH, Recklinghausen
  - Uniklinikum Ulm, Klinik für Innere Medizin II, Pneumologie, Ulm

REFERENCES:
- [Derived] Schuette W, Behringer D, Stoehlmacher J, Kollmeier J, Schmager S, Fischer von Weikersthal L, Schumann C, Buchmann J. CHAMP: A Phase II Study of Panitumumab With Pemetrexed and Cisplatin Versus Pemetrexed and Cisplatin in the Treatment of Patients With Advanced-Stage Primary Nonsquamous Non-Small-Cell Lung Cancer With Particular Regard to the KRAS Status. Clin Lung Cancer. 2015 Nov;16(6):447-56. doi: 10.1016/j.cllc.2015.05.009. Epub 2015 Jun 2. PMID 26094080